CLINICAL TRIAL: NCT00493259
Title: Health-related Quality of Life, Depression and the Impact on Successful Incorporation of Lifestyle Changes in Insulin Resistant Adolescents as Evidenced by Changes in BMI, Waist Circumference and Metabolic Parameters
Brief Title: Health Related QOL, Depression and Lifestyle Changes in Insulin Resistant Adolescents
Status: Completed | Type: Observational
Sponsor: Children's Mercy Hospital Kansas City (Other)
Responsible Party: Sponsor
Other Study IDs: 07 02-037E
Record Dates: First submitted 2007-06-26; First posted 2007-06-28 (Estimated); Last update posted 2021-01-06 (Actual); Status verified 2021-01

CONDITIONS: Insulin Resistance; Depression
Keywords: Health-Related Quality of Life
MeSH Terms: conditions — Insulin Resistance; Depression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: Health-Related Quality of Life instrument — Adolescents will fill out questionnaires regarding quality of life and dealing with diagnosis of Insulin Resistance Syndrome
Behavioral: Depression Scale for Children (CES-DC) — questionnaire

SUMMARY:
The purpose of this study is to assess adolescents with Insulin Resistance Syndrome for quality of life and altered health related issues.

DETAILED DESCRIPTION:
Matched historical control study designed to examine outcomes on insulin resistant adolescents who were treated in the Insulin Resistance Syndrome Clinic at Children's Mercy Hospital in the past year. New patients will be screened at baseline, 4 and 12 months to evaluate if there is improvement in the BMI Z-score, HgA1c, lipid profile or waist circumference when depression and/or altered health related quality of life are identified and treated in this population.

ELIGIBILITY:
Inclusion Criteria:

* Patients 11-17 years of age who are seen in the Insulin Resistance Clinic for the first time
* Historical control: Patients 11-19 years of age seen in the Insulin Resistance Clinic during the prior four months

Exclusion Criteria:

* Co-morbid syndrome (Downs, Turner's, Prader Willi etc)
* Diagnosis of Type 2 Diabetes
* Taking Metformin before the initial visit
* Taking medication for or diagnosis of a psychiatric condition prior to initial visit
* Developmentally delayed

Ages: 11 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adoslescents treated in Children's Mercy Hospital and Clinic, Endocrine clinic.
Sampling Method: Non-Probability Sample
Enrollment: 78 (Actual)
Dates: Start 2007-06 (Actual); Primary Completion 2008-06 (Actual); Study Completion 2008-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Adrienne Platt, MS, CPNP, Principal Investigator — Children's Mercy Hospital Kansas City
Locations (1):
- Children's Mercy Hospital, Kansas City, Missouri, United States